CLINICAL TRIAL: NCT00570414
Title: Airway Management in Children Undergoing Adenotonsillectomies Under General Anesthesia; a Comparison of the Endotracheal Tube and the Laryngeal Mask Airway
Brief Title: Airway Management in Children Undergoing Adenotonsillectomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Telemark (Other Government)
Responsible Party: Simen Doksrød, Sykehuset Telemark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: s8197.03; s-07031b
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Last update posted 2009-01-15 (Estimated); Status verified 2009-01

CONDITIONS: Tonsillitis
MeSH Terms: conditions — Tonsillitis | interventions — Laryngeal Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Laryngeal mask airway (LMA)
  Interventions: Device: Laryngeal mask airway
- 2 (Active Comparator): Endotracheal tube (ETT)
  Interventions: Device: Endotracheal tube

INTERVENTIONS:
Device: Laryngeal mask airway — Airway management by the use of the flexible, reinforced laryngeal mask airway
  Arms: 1
Device: Endotracheal tube — Airway management by the use of endotracheal tube
  Arms: 2

SUMMARY:
Secure airway management is the basis of all anesthesiological practice. Of particular importance is the securing of patients' airway passages when the surgical procedure itself poses a threat to a patient's airway, as is the case in all procedures involving the upper respiratory pathways. When adenoidectomies, tonsillectomies and combined adenotonsillectomies are performed, blood from the surgical area will present a respiratory threat to unsecured airways. The traditional opinion has been that endotracheal intubation is the safest method of preventing aspiration.

The laryngeal mask was introduced in 1983 as an alternative to the endotracheal tube. In 1990, the flexible, reinforced laryngeal mask airway was introduced, intended for use during surgical procedures involving the mouth and throat. The laryngeal mask airway has several potential advantages over the endotracheal tube. It is inserted blindly, without laryngoscopy. This leads to reduced oropharyngeal or laryngeal stimulation and injury, and therefore minimal activation of respiratory and circulatory reflexes. The laryngeal mask airway can be placed without the use of muscle relaxants, avoiding potential side effects such as apnea, hyperkalemia and anaphylaxis. In addition the laryngeal mask airway can remain in the throat until the patient awakes, virtually eliminating the danger of postoperative aspiration.

Several international studies have described the advantages of the laryngeal mask airway over endotracheal intubation during ear, nose and throat surgery in children. The general impression is that there is a widespread routine implementation of the laryngeal mask airway. In Norway, however, this practice has been limited. As far as we know, only Namsos Hospital uses this procedure as its first choice. At Telemark Hospital we tested the use of laryngeal mask airway on 150 patients between May and December 2006. The results so far have been promising, and we have had no serious complications.

Hypothesis:

In children undergoing adenotonsillectomies, a laryngeal mask airway provides greater patient satisfaction (judged by reduced pain, nausea and vomiting) and greater effectivity (judged by reduced time in surgery), compared with the endotracheal tube. The laryngeal mask provides as much as or greater secure airway management measured by desaturations/Sp02<92% and/or use of suxamethonium and bronchiolytic drugs.

DETAILED DESCRIPTION:
Registration:

Preoperative: Age, height, weight, medication, asthma/allergy, possible current respiratory infection

Peroperative: Type of procedure, tube size/laryngeal mask, type of tongue blade, highest/lowest SpO2, highest/lowest ET CO2, highest/lowest pulse, length of surgery, total operating room time, operator, medication. Reason must be given if converting from laryngeal mask to tube; lack of visibility for operator, laryngeal mask not possible to place, unacceptable leakage before placing tongue blade, occlusion after placement of tongue blade.

Postoperative: Pain judged by need for opiates (VAS, crying, agitation, tachycardia), nausea judged by gagging/vomiting, total time in recovery, rebleeding judged by reoperation.

Anesthesia:

Induction: Alfentanil 20 microg/kg body weight Propofol 3-4 mg/kg body weight Or: Sevoflurane/N2O mask induction with MAC 1-2

Maintenance: Alfentanil 5-10 microg/kg body weight every 8-10 minutes Sevoflurane/N2O equivalent to 1-1.5 MAC Acetaminophen supp 40 mg/kg body weight, max 2 g. Dexamethasone 0.15mg/kg body weight Xylocaine 1mg/kg body weight

Emergence: Morphine 100-200 mikrog/kg body weight

Postoperative: Morphine 50-100 microg/kg body weight

Post-discharge: Acetaminophen tbl 15 mg/kg body weight x 3 Or: Acetaminophen supp 20 mg/kg body weight x 3

Patient booklet:

A patient booklet will be produced for each patient. The booklet will contain only the patient's initials, age and research number. After the booklets are filled out, they will be stored in a locked facility by one of the examining physicians, and the code to the patient's name will be stored and locked separately by one of the researchers. The code will be destroyed at the end of the research study.

ELIGIBILITY:
Inclusion Criteria:

* Children 10-60 kg
* Elective adenotomy, tonsillectomy or combined adenotonsillectomy under general anesthesia.
* Written and oral informed parental consent.

Exclusion Criteria:

* ASA III or higher.
* Weight < 10 kg or weight > 60 kg.
* Congenital malformations of the mouth or throat.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2007-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction: a) Pain (VAS, use of opioids), b) Nausea and vomiting (score) | 24 hrs

SECONDARY OUTCOMES:
Effectivity (judged by reduced time in surgery) | 1 hrs
Secure airway management measured by desaturations/Sp02<92% and/or use of suxamethonium and bronchiolytic drugs. | 24 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Simen Doksrød, MD, Principal Investigator — Sykehuset Telemark; Peter Heidt, PhD, Study Director — Namsos Hospital
Locations (1):
- Sykehuset Telemark, Clinic of emergency medicin, Porsgrunn, Telemark, Norway